CLINICAL TRIAL: NCT03536910
Title: Evaluation of Copeptin Levels in Elective Cesarean Section With Spinal and General Anesthesia and Their Relationship With Fetal Stress: Prospective Study
Brief Title: Evaluation of Copeptin Levels in Elective Cesarean Section With Different Anesthetic Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Ece YAMAK ALTINPULLUK, Principal Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: No protocol ID
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Fetal Distress
Keywords: copeptin levels; Cesarean section; general anesthesia; spinal anesthesia
MeSH Terms: conditions — Fetal Distress | interventions — Arginine Vasopressin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General anesthesia (Other)
  Interventions: Other: Copeptin
- Spinal anesthesia (Other)
  Interventions: Other: Copeptin

INTERVENTIONS:
Other: Copeptin — Level of copeptin in maternal blood and umbilical cord blood
  Other Names: Fetal distress

SUMMARY:
In this study, investigators aimed to investigate the effects of general and spinal anesthesia techniques on copeptin levels during cesarean section and their relation with fetal distress.

DETAILED DESCRIPTION:
During the delivery process, the mother and the baby generate some endocrine responses to this emotional and physical stressful action. Arginin-Vasopressin prohormone (copeptin), which is more stable and measurable in blood, is used as an endogenous stress indicator. Copeptin levels have been shown to be significantly increased in vaginally delivery when compared to cesarean section (c / s). In a caesarean section; it is a known fact that when the general anesthetic method and the used anesthetic substances are taken into consideration, it gives a significant stress to the mother and the baby. Spinal anesthesia with no impaired fetal oxygenation and without orotracheal intubation and neuromuscular blockers may reduce fetal distress. However, there was no study investigating the effect of the anesthesia techniques in elective cesarean section on the fetal stress and the level of copeptin, in the literature review. Therefore investigators aimed to compare spinal and general anesthesia technique in elective cesarean section, to evaluate level of copeptin and their relation with fetal distress.Investigators hope that this study will guide the anesthesia method that can be chosen primarily in caesarean section.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years of age
* ASA I-II
* 36-40 gestational weeks
* BMI ≤ 40
* Undergoing elective cesarean section

Exclusion Criteria:

* Coagulopathy
* Known central or peripheral nerve disease
* fetal anomalies
* birth weight less than 2000 grams and above 4500 grams,
* infants with a risk of meconium or amniotic fluid aspiration
* kidney failure, diabetes mellitus, hypertension, cardiac disease, antepartum hemorrhage, asthma bronchiole, Rh incompatibility, congenital malformations

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnancy
Enrollment: 60 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Changes in copeptin levels after general or spinal anesthesia | Baseline and immediately after surgery from maternal blood and arterial and venous umbilical cord at birth

CONTACTS AND LOCATIONS:
Overall Officials: Ece YAMAK ALTINPULLUK, MD, Principal Investigator — Istanbul University
Locations (1):
- Istanbul University Cerrahpasa Medical Faculty, Istanbul, Turkey (Türkiye)